CLINICAL TRIAL: NCT06423066
Title: Developing a Machine Learning Model to Predict Pleural Adhesion Preoperatively Using Pleural Ultrasound: a Prospective Observational Study
Brief Title: Developing a Machine Learning Model to Predict Pleural Adhesion Preoperatively Using Pleural Ultrasound
Status: Not yet recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Xuehan Gao, Research Investigator, Peking Union Medical College Hospital
Other Study IDs: USPDPA01
Record Dates: First submitted 2024-05-15; First posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Pleural Diseases; Lung Cancer; Machine Learning
Keywords: pleural adhesion; 3D-CNN; machine learning; VATS
MeSH Terms: conditions — Pleural Diseases; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pleural ultrasound group: Patients who accept pleural ultrasound preoperatively.
  Interventions: Diagnostic Test: Pleural ultrasound

INTERVENTIONS:
Diagnostic Test: Pleural ultrasound — Patients who examine pleural ultrasound preoperatively.

SUMMARY:
This study aims to investigate the accuracy of using pleural ultrasound (USP) to identify pleural adhesions in patients who plan to receive video-assisted thoracoscopic surgery. It employs three-dimensional convolutional neural network (3D-CNN) technology to process USP-related images and video data for machine learning, and to establish a diagnostic model for identifying pleural adhesions using 3D-CNN-USP. The study will determine the sensitivity, specificity, positive predictive value, and negative predictive value of 3D-CNN-USP in identifying pleural adhesions. Additionally, it will explore the feasibility and effectiveness of using 3D-CNN-USP for preoperative identification of pleural adhesions in VATS, thereby supporting the implementation of day surgery in thoracic surgery and ultimately serving clinical practice.

DETAILED DESCRIPTION:
Lung cancer is currently the leading cause of death from malignant tumors worldwide. Surgery is the primary treatment method for lung cancer, and breakthroughs in thoracic surgical techniques play a crucial role in the diagnosis and treatment of lung cancer. Medical ultrasound technology, due to its non-invasive, flexible, convenient, and economical characteristics, is widely used in clinical practice. With the advancement of ultrasound technology and the need to address clinical challenges, ultrasound imaging technology has seen new developments in the field of thoracoscopic surgery.

In the era of minimally invasive surgery, intraoperative pleural adhesions are one of the main factors affecting the implementation of video-assisted thoracoscopic surgery (VATS). Especially under the concept of enhanced recovery after surgery (ERAS), the day surgery model for VATS has gradually taken shape. However, pleural adhesions significantly increase intraoperative trauma and prolong hospital stays. Additionally, pleural adhesions increase the risk of lung injury during VATS and, in severe cases, may hinder access to the pleural space, necessitating conversion to open thoracotomy. Pleural adhesions increase intraoperative time and morbidity in thoracic surgery due to poor visibility, bleeding, and lung and vascular injuries. The presence, location, and degree of pleural adhesions are useful for determining the initial port placement or choosing between open or VATS approaches. Therefore, accurately predicting the presence and specific location of pleural adhesions preoperatively is crucial for the development of day surgery under thoracic ERAS, ensuring the safety and efficiency of future VATS day surgeries.

Previous studies have shown that chest CT is difficult to predict pleural adhesions, with a sensitivity of only 72% and a sensitivity of only 46% for determining adhesions at specific locations. In contrast, ultrasonography of the pleura (USP) can dynamically display pleural sliding and adhesions with surrounding lung tissue, and has real-time monitoring capabilities based on movement, providing unique advantages for detecting pleural adhesions. Preoperative prediction of pleural adhesions using USP has significant application value. Studies have already demonstrated the advantages of using transthoracic pleural ultrasound to identify pleural adhesions. Nicola et al. conducted 1,192 ultrasounds to predict pleural adhesions, confirming 1,124 positive cases and 68 negative cases, with a sensitivity of 80.6%, specificity of 96.1%, positive predictive value of 73.2%, and negative predictive value of 97.4%. However, there are still some issues with using USP to predict pleural adhesions. Physicians who can identify pleural adhesions need to be trained in lung ultrasound, and ultrasound examination and interpretation are skill-dependent techniques. The burden of training thoracic ultrasound physicians remains a clinical challenge.

Three-dimensional convolutional neural network (3D-CNN) technology is an emerging technology in the field of artificial intelligence and machine learning. Unlike traditional convolutional neural networks (CNN), 3D-CNN can process three-dimensional data that includes a time dimension, making it suitable for analyzing the real-time dynamic image features of ultrasound images. This technology holds promise for developing a machine learning model to interpret USP images, potentially replacing physician interpretation and improving the accuracy of USP in identifying pleural adhesions.

In summary, this study intends to use USP for preoperative identification of pleural adhesions in patients scheduled for VATS surgery. It aims to investigate the accuracy of USP in predicting intraoperative pleural adhesions and to develop a diagnostic model using 3D-CNN technology to process USP-related images and video data for machine learning. The study will explore the sensitivity, specificity, positive predictive value, and negative predictive value of the 3D-CNN-USP model in identifying pleural adhesions. Additionally, it will examine the feasibility and effectiveness of using 3D-CNN-USP for preoperative identification of pleural adhesions to support the implementation of day surgery in thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who plan to accept VATS surgery.

Exclusion Criteria:

1. Patients who can not obtain detailed clinical information;
2. Patients or their family members who can not understand the conditions and objectives of the study or refuse to participate in the study;
3. Patients with conditions affecting observation, such as skin lesions, infections, or scars in the area of the chest wall to be examined.

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who plan to accept VATS surgery in Peking Union Medical college Hospital, and agree to perform preoperative plerual ultrasound examination.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | From enrollment to the end of surgery.
  Sensitivity of three-dimensional convolutional neural network (3D-CNN) in identifying pleural adhesions using pleural ultrasound (USP). The sensitivity value ranges from 0 to 100, with higher values indicating greater sensitivity.

SECONDARY OUTCOMES:
Specificity | From enrollment to the end of surgery.
  Specificity off 3D-CNN in identifying pleural adhesions using USP. The specificity value ranges from 0 to 100, with higher values indicating greater specificity.
Positive predictive value | From enrollment to the end of surgery.
  Positive predictive value (PPV) of 3D-CNN in identifying pleural adhesions using USP. PPV is calculated by dividing the number of true positive results by the total number of positive test results. A higher PPV means that the test is more reliable in correctly identifying those with the condition.
Negative predictive value | From enrollment to the end of surgery.
  Negative predictive value (NPV) of 3D-CNN in identifying pleural adhesions using USP. NPV is calculated by dividing the number of true negative results by the total number of negative test results. A higher NPV means that the test is more reliable in correctly identifying those without the condition.

CONTACTS AND LOCATIONS:
Overall Officials: Shanqing Li, PhD, and MD, Study Director — Peking Union Medical College Hospital; Qingli Zhu, PhD, and MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The data of this study will be used in future analyses and be published in academic article.

REFERENCES:
- [Background] Mason AC, Miller BH, Krasna MJ, White CS. Accuracy of CT for the detection of pleural adhesions: correlation with video-assisted thoracoscopic surgery. Chest. 1999 Feb;115(2):423-7. doi: 10.1378/chest.115.2.423. PMID 10027442
- [Background] Cassanelli N, Caroli G, Dolci G, Dell'Amore A, Luciano G, Bini A, Stella F. Accuracy of transthoracic ultrasound for the detection of pleural adhesions. Eur J Cardiothorac Surg. 2012 Nov;42(5):813-8; discussion 818. doi: 10.1093/ejcts/ezs144. Epub 2012 Apr 19. PMID 22518039